CLINICAL TRIAL: NCT01835041
Title: A Phase I Open-Label Dose-Escalation Clinical Trial of CPI-613 in Combination With Modified FOLFIRINOX in Patients With Metastatic Pancreatic Cancer and Good Performance Status
Brief Title: CPI-613 and Combination Chemotherapy in Treating Patients With Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00022532; NCI-2013-00674 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA012197 (NIH); CCCWFU 57112 (Other: Wake Forest Baptist Comprehensive Cancer Center)
Record Dates: First submitted 2013-04-16; First posted 2013-04-18 (Estimated); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Acinar Cell Adenocarcinoma of the Pancreas; Duct Cell Adenocarcinoma of the Pancreas; Recurrent Pancreatic Cancer; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — devimistat; Oxaliplatin; Leucovorin; Irinotecan; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (6,8-bis[benzylthio]octanoic acid, mFOLFIRINOX) (Experimental): Patients receive 6,8-bis(benzylthio)octanoic acid IV over 2 hours on days 1 and 3. Patients also receive oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, irinotecan hydrochloride IV over 90 minutes, and fluorouracil IV continuously over 46 hours on day 1. Treatment repeats every 2 weeks for 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: 6,8-bis(benzylthio)octanoic acid; Drug: oxaliplatin; Drug: leucovorin calcium; Drug: irinotecan hydrochloride; Drug: fluorouracil; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: 6,8-bis(benzylthio)octanoic acid — Given IV
  Other Names: alpha-lipoic acid analogue CPI-613; CPI-613
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
Drug: leucovorin calcium — Given IV
  Other Names: CF; CFR; LV
Drug: irinotecan hydrochloride — Given IV
  Other Names: Campto; Camptosar; CPT-11; irinotecan; U-101440E
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of CPI-613 when given together with combination chemotherapy in treating patients with metastatic pancreatic cancer. Drugs used in chemotherapy, CPI-613, leucovorin calcium, fluorouracil, irinotecan hydrochloride, and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of CPI-613 (6,8-bis[benzylthio]octanoic acid), when used in combination with modified leucovorin calcium, fluorouracil, irinotecan hydrochloride, and oxaliplatin (mFOLFIRINOX), in patients with metastatic pancreatic cancer.

SECONDARY OBJECTIVES:

I. To assess the safety of CPI-613/mFOLFIRINOX combination in patients with metastatic pancreatic cancer.

II. To collect tissue for future genomic analyses. III. To obtain preliminary data on efficacy of treatment with CPI-613/mFOLFIRINOX.

OUTLINE: This is a dose-escalation study of 6,8-bis(benzylthio)octanoic acid.

Patients receive 6,8-bis(benzylthio)octanoic acid intravenously (IV) over 2 hours on days 1 and 3. Patients also receive oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, irinotecan hydrochloride IV over 90 minutes, and fluorouracil IV continuously over 46 hours on day 1. Treatment repeats every 2 weeks for 6 months in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically and cytologically confirmed metastatic pancreatic adenocarcinoma
* Eastern Cooperative Oncology Group (ECOG) performance status being 0-1
* Expected survival > 2 months
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must use accepted contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive or double barrier device) during the study, and must have a negative serum or urine pregnancy test within 1 week prior to treatment initiation
* Fertile men must practice effective contraceptive methods during the study, unless documentation of infertility exists
* At least 2 weeks must have elapsed from any prior surgery or hormonal therapy
* Granulocyte count >= 1500/mm^3
* White blood cell (WBC) >= 3500 cells/mm^3 or >= 3.5 bil/L
* Platelet count >= 100,000 cells/mm^3 or >= 100 bil/L
* Absolute neutrophil count (ANC) >= 1500 cells/mm^3 or >= 1.5 bil/L
* Hemoglobin >= 9 g/dL or >= 90 g/L
* Aspartate aminotransferase (AST/serum glutamic oxalic transaminase [SGOT]) =< 3 x upper normal limit (UNL), alanine aminotransferase (ALT/serum glutamate pyruvate transaminase [SGPT]) =< 3 x UNL (=< 5 x UNL if liver metastases present)
* Bilirubin =< 1.5 x UNL
* Serum creatinine =< 2.0 mg/dL or 177 µmol/L
* International normalized ratio or INR must be =< 1.5 unless on therapeutic blood thinners
* No evidence of active infection and no serious infection within the past month
* Mentally competent, ability to understand and willingness to sign the informed consent form

Exclusion Criteria:

* Endocrine or acinar pancreatic carcinoma
* Previous radiotherapy for cerebral metastases, central nervous system (CNS) or epidural tumor
* Prior treatment with any chemotherapy for metastatic disease from pancreatic cancer
* Patients receiving any other standard or investigational treatment for their cancer, or any other investigational agent for any indication within the past 4 weeks prior to initiation of CPI-613 treatment
* Serious medical illness that would potentially increase patients' risk for toxicity
* Any active uncontrolled bleeding, and any patients with a bleeding diathesis (e.g., active peptic ulcer disease)
* Pregnant women, or women of child-bearing potential not using reliable means of contraception (because the teratogenic potential of CPI-613 is unknown)
* Lactating females
* Fertile men unwilling to practice contraceptive methods during the study period
* Life expectancy less than 2 months
* Any condition or abnormality which may, in the opinion of the investigator, compromise the safety of patients
* Unwilling or unable to follow protocol requirements
* Active heart disease including but not limited to symptomatic congestive heart failure, symptomatic coronary artery disease, symptomatic angina pectoris, symptomatic myocardial infarction, or symptomatic congestive heart failure
* Patients with a history of myocardial infarction that is < 3 months prior to registration
* Evidence of active infection, or serious infection within the past month
* Patients with known human immunodeficiency virus (HIV) infection
* Patients who have received immunotherapy of any type within the past 4 weeks prior to initiation of CPI-613 treatment
* Requirement for immediate palliative treatment of any kind including surgery
* Patients that have received a chemotherapy regimen with stem cell support in the previous 6 months
* Any condition or abnormality which may, in the opinion of the investigator, compromise the safety of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2023-03-16 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 2 weeks
  of 6,8-bis(benzylthio)octanoic acid when used in combination with mFOLFIRINOX determined by dose-limiting toxicities graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.0

OTHER OUTCOMES:
Number of Toxicities | Approximately 2 month after start of treatment or completion of Cycle 2
  For exploratory purposes - Any toxicities greater than Grade 2 or above will be assessed for safety of use of CPI-613 and mFOLFIRINOX.
Overall Survival | Approximately 6 months after start of treatment
  For exploratory purposes - Overall survival curve will be measured using Kaplan-Meier methods. Medial survival rates will be examined using a 95% confidence interval.
Progression-Free Survival | Approximately 2 months after start of treatment
  For exploratory purposes - The duration of clinical response (evaluated by progression free survival) will be measured from the date a first objective response is documented until the first sign of progression assessed by MRI.
Number of Participants with a Clinical Response | Approximately 2 months after start of treatment
  For exploratory purposes - CA-19-9 will be collected every fourth cycle along with MRI of the abdomen and contrast CT of the chest for clinical response.

CONTACTS AND LOCATIONS:
Overall Officials: Caio Rocha Lima, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States

REFERENCES:
- [Derived] Liu N, Yan M, Tao Q, Wu J, Chen J, Chen X, Peng C. Inhibition of TCA cycle improves the anti-PD-1 immunotherapy efficacy in melanoma cells via ATF3-mediated PD-L1 expression and glycolysis. J Immunother Cancer. 2023 Sep;11(9):e007146. doi: 10.1136/jitc-2023-007146. PMID 37678921
- [Derived] Alistar A, Morris BB, Desnoyer R, Klepin HD, Hosseinzadeh K, Clark C, Cameron A, Leyendecker J, D'Agostino R Jr, Topaloglu U, Boteju LW, Boteju AR, Shorr R, Zachar Z, Bingham PM, Ahmed T, Crane S, Shah R, Migliano JJ, Pardee TS, Miller L, Hawkins G, Jin G, Zhang W, Pasche B. Safety and tolerability of the first-in-class agent CPI-613 in combination with modified FOLFIRINOX in patients with metastatic pancreatic cancer: a single-centre, open-label, dose-escalation, phase 1 trial. Lancet Oncol. 2017 Jun;18(6):770-778. doi: 10.1016/S1470-2045(17)30314-5. Epub 2017 May 8. PMID 28495639

DOCUMENTS (1):
  • Informed Consent Form (2021-05-18): https://cdn.clinicaltrials.gov/large-docs/41/NCT01835041/ICF_000.pdf